CLINICAL TRIAL: NCT01806051
Title: A Pilot Study on the Diurnal Variation in PKU Patients With Kuvan
Brief Title: A Pilot Study on Diurnal Variation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participants found the study procedures to be too cumbersome and no longer wanted to participate
Sponsor: Dr. Linda Randolph (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Dr. Linda Randolph, Head, Division of Medical Genetics, Children's Hospital Los Angeles
Organization: Children's Hospital Los Angeles (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CCI-12-00178
Record Dates: First submitted 2013-03-04; First posted 2013-03-07 (Estimated); Results first posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-03

CONDITIONS: Phenylketonuria (PKU)
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PKU Participants (Arm 1) (Experimental): * Subjects will be administered Kuvan once daily.
  * They will undergo several blood draws, including a 24-Hour Blood Assessment (at Study Visit #2 before the commencement of Kuvan), plasma Phe/Tyr draws (at Study Visits #3, 4, and 5), and another 24-Hour Blood Assessment (at Study Visit #6).
  Interventions: Drug: Kuvan
- Control Group (Arm 2) (No Intervention): * Subjects allocated into this group will be healthy, non-PKU individuals that may be a relative (ex: sibling) of a PKU participant, but they don't have to be a blood relation.
  * These subjects will undergo a 24-Hour Blood Assessment (at Study Visit #2).

INTERVENTIONS:
Drug: Kuvan — Only PKU participants (Arm 1) will be administered Kuvan once daily either at a dose of 20 mg/kg/day (if the PKU participant is not currently taking Kuvan) or at the subject's regular dose (if the PKU participant is currently taking Kuvan). They will remain on Kuvan for 4 weeks.
  Arms: PKU Participants (Arm 1)

SUMMARY:
This self-controlled, prospective, pilot study is designed to gather information regarding the diurnal variation (changes that occur each day) in the levels of plasma phenylalanine (Phe) and tyrosine in patients with phenylketonuria (PKU) and in the non-PKU population.

DETAILED DESCRIPTION:
Phenylketonuria (PKU) is a rare genetic metabolic disease caused by a mutation that codes for an enzyme that converts the essential amino acid phenylalanine (Phe) into tyrosine. An absence or deficiency of this enzyme activity results in a Phe elevation, where higher Phe levels result in neurological damage. Diurnal variations of Phe levels have been observed in PKU patients in a 24-hour period.

As Kuvan has shown to stabilize Phe levels in PKU patients over time, our hypothesis is that this can be demonstrated within a 24-hour period of observation and indicate therefore that Kuvan may correlate with a lower plasma Phe variability. This study on PKU patients' diurnal variation will also provide important information as to the current method of blood Phe monitoring in a clinical setting to learn more about the optimal way to measure Phe concentration.

The study will last about 4 weeks (6 study visits) for the PKU participants and about 1 week (2 study visits) for the control group.

Participants will be required to follow a recommended diet, complete a dietary log, and undergo several blood draws, including a 24-Hour Blood Assessment in which blood will be obtained 8 times throughout the day.

ELIGIBILITY:
Inclusion Criteria:

PKU PARTICIPANTS (ARM 1):

* Subject has a confirmed diagnosis of PKU with hyperphenylalaninemia documented by a fasting Phenylalanine level of at least 360 umol/L (6 mg/dL)
* Patient is at least 4 years old (there is no upper age limit for this study)
* Willing and able to provide written authorization or, if under the age of 18 years, provide written assent (if required) and written patient authorization by a parent or legal guardian
* Willing to undergo study related procedures including commencing Kuvan treatment for patient not currently on treatment; temporary discontinuation of Kuvan for patient on treatment; and completing the 24-Hour Blood Assessment
* Authorized to provide personal health information
* Subjects should not be pregnant and willing to use appropriate birth control during the study

CONTROL GROUP (ARM 2):

* Healthy, non-PKU individuals. They will be age-sex matched to the PKU group. They may be a relative (ex: sibling) of a PKU participant, but they don't have to be a blood relation.
* Individual is at least 4 years old (there is no upper age limit)
* Willing and able to provide written consent or, if under the age of 18 years, provide written assent and written participant authorization by a parent or legal guardian
* Authorized to provide personal health information

Exclusion Criteria (BOTH ARMS):

* Subjects who do not meet all the inclusion criteria
* Age < 4 years
* Concomitant medical problems or medications which at the discretion of the principal investigator would put participant at health risk or prevent them from completing study.
* If female, unwillingness to use birth control during the period of the study drug administration (this doesn't apply to Arm 2)

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda M. Randolph, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No data was collected because all of the participants who consented to participate in the study withdrew due to the procedural challenges of remaining in the study (e.g. the PM blood draws were too disruptive).
Groups:
- All Participants: Participants signed the consent forms and withdrew because they found the study procedures to be too cumbersome.
Period: Overall Study
Arm/Group | All Participants
Started | 6
Completed | 0
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Population: Participants withdrew before baseline characteristics were collected.
Arm/Group | All Participants
Number analyzed (Participants) | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Changes in Plasma Phe and Tyrosine Levels
Description: To evaluate the patterns of change in plasma Phe and tyrosine levels between the Baseline visit and 4 week visit for each arm.
Time Frame: Baseline and 4 weeks
Population: Participants withdrew before any data were collected.
Groups:
- PKU Participants (Arm 1): * Subjects will be administered Kuvan once daily.
  * They will undergo several blood draws, including a 24-Hour Blood Assessment (at Study Visit #2 before the commencement of Kuvan), plasma Phe/Tyr draws (at Study Visits #3, 4, and 5), and another 24-Hour Blood Assessment (at Study Visit #6).
  Kuvan: Only PKU participants (Arm 1) will be administered Kuvan once daily either at a dose of 20 mg/kg/day (if the PKU participant is not currently taking Kuvan) or at the subject's regular dose (if the PKU participant is currently taking Kuvan). They will remain on Kuvan for 4 weeks.
Arm/Group | PKU Participants (Arm 1) | Control Group (Arm 2)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Participants withdrew before any data were collected.
Arm/Group | PKU Participants (Arm 1) | Control Group (Arm 2)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No